CLINICAL TRIAL: NCT04572464
Title: A Pre-Experimental Study to Assess the Effectiveness of Mindfulness Based Guided Meditation on Wellbeing, Self Compassion and Cognizance Among Nurses Working in Intensive Care Units at ILBS, New Delhi
Brief Title: Effectiveness of Mindfulness Based Meditation on Well-being, Self Compassion & Cognizance Among Nurses Working in Intensive Care Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: F15(2/2.25)/2017/HO(M)/ILBS
Record Dates: First submitted 2020-07-22; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2019-11

CONDITIONS: Mindfulness is a Moment by Moment Awareness to Remain Purposefully and Non Judgmentally Attentive to Their Own Experience

STUDY DESIGN:
Intervention Model Description: One group pre test post test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Mindfulness Based Guided Meditation
  Interventions: Other: Mindfulness Based Guided Meditation

INTERVENTIONS:
Other: Mindfulness Based Guided Meditation — Mindfulness Based Guided Meditation will be practiced by nurses under the supervision of researcher for 15 min thrice a week for two weeks

SUMMARY:
Effect of Mindfulness Based Guided Meditation on Intensive care Unit nurses wellbeing,cognizance & self compassion was assessed .

DETAILED DESCRIPTION:
: Primary objective To assess the Effectiveness of Mindfulness Based Guided Meditation on Wellbeing, Self Compassion and Cognizance among Nurses working in Intensive Care Units at ILBS.

Hypothesis

The following hypothesis will be tested at 0.05 level of significance:

H1There will be a significant difference between pretest Wellbeing scores and posttest Wellbeing scores of Nurses working in Intensive Care Units. H2There will be a significant difference between pretest Self Compassion Scores and posttest Self Compassion scores of Nurses working in Intensive Care Unit.

H3There will be a significant difference between pretest Cognizance Scores and posttest Cognizance score of Nurses Working in Intensive Care Units.

H4 There will be a significant relationship between Wellbeing and Self Compassion Among Nurses working in Intensive Care Units.

H5 There will be a significant relationship between Wellbeing and Cognizance among Nurses working in Intensive Care Units.

H6 There will be a significant relationship between Self Compassion and Cognizance Among Nurses working in Intensive Care Units.

H7 There will be a significant association of posttest wellbeing score with selected Socio demographic variables of Nurses working in Intensive Care Units.

H8 There will be a significant association of posttest Self Compassion score with selected sociodemographic variables of Nurses working in Intensive Care Units.

H9 There will be a significant association of Posttest Cognizance score with selected sociodemographic variables of Nurses working in Intensive Care Units.

Research Design Pre-experimental, one group pre test -post test design

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses who were Working in ICUs for at least last three months continuously.

Exclusion Criteria:

* Registered nurses who were On long leave Had joined recently in ICUs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Wellbeing | 10 minutes
  The study will be carried out among Nurses working in Intensive Care Units at ILBS Hospital using Total enumeration technique. The primary outcome measure will be increase in post test wellbeing scores among nurses as compared to their pretest wellbeing scores which will be assessed by using Warwick Edinburgh Mental Wellbeing scale in about 10 mins.
Self Compassion | 15 minutes
  The study will be carried out among Nurses working in Intensive Care Units at ILBS hospital using Total enumeration technique.The primary outcome measure will be increase in post test Self Compassion scores among nurses as compared to their pre test Self Compassion scores which will be measured using Self Compassion Scale in about 15 mins.
Self Compassion | 10 minutes
  The study will be carried out among Nurses working in Intensive Care Units at ILBS hospital using Total enumeration technique. The primary outcome measure will be increase in post test Cognizance score among nurses as compared to their pretest Cognizance scores which will be measured using Mindful Attention Awareness Scale in about 10 mins

CONTACTS AND LOCATIONS:
Locations (1):
- Neetu Taneja, Faridabad, Haryana, India